CLINICAL TRIAL: NCT00035399
Title: Efficacy of Acupuncture With Physical Therapy for Knee Osteo-Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: John T. Farrar, MD, PhD, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000304-01A1 (NIH)
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Osteoarthritis
Keywords: acupressure /acupuncture; alternative medicine; arthritis therapy; combination therapy; human therapy evaluation; knee; osteoarthritis; physical therapy; chronic pain; clinical trial; functional ability
MeSH Terms: conditions — Osteoarthritis; Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
This study will examine the efficacy of acupuncture in combination with exercise physical therapy for moderate osteoarthritis (OA) of the knee.

DETAILED DESCRIPTION:
Acupuncture is an ancient Chinese technique of using a fine needle to stimulate points along theoretical meridians of energy to correct imbalances thought to be responsible for specific disease states. In the United States, acupuncture is often used for the treatment of painful conditions. The 1997 NIH Consensus Conference concluded that there was adequate evidence of efficacy in an acute dental pain model and in nausea. In chronic pain, most studies were too small, poorly designed, poorly executed, or improperly controlled to adequately demonstrate that needle acupuncture worked better than sham acupuncture, placebo, standard medical therapy, or even no treatment. Osteoarthritis (OA) of the knee has been proposed as a good model to test the efficacy of acupuncture in a chronic pain condition because it is an extremely common, well defined, and disabling condition with well established outcome measures for symptoms and functional status. There is clinical trial evidence of efficacy for the standard treatments of acetaminophen and NSAIDs, and exercise physical therapy (EPT), which is usually added when the patient develops functional limitations. One high quality study of acupuncture for knee OA, demonstrated moderate benefit in an unblinded comparison to a usual care control group. As such, a major question remains about whether acupuncture, used in addition to exercise therapy, will provide a clinically meaningful improvement in pain and function. Since pain can be the primary limiting factor in improved exercise capacity, if acupuncture has any efficacy in reducing the pain of knee OA, then the combination with an EPT program should be substantially more effective than EPT alone. Another major concern is that the effect of the acupuncture may be predominantly mediated by non- specific placebo effects rather than the specific effects of the placement of a needle. Another important component of this proposal is our use of a validated blinded placebo needle instead of sham acupuncture points. Therefore, the primary goal of this proposal is to use a properly designed randomized blinded clinical trial, using American College of Rheumatology (ACR) criteria and Food and Drug Administration (FDA) recommended outcome measures, to determine whether the addition of acupuncture to standard EPT provides an overall clinically important benefit to patients with symptomatic knee OA compared to placebo acupuncture. As a secondary goal, we will use the clinical trial data to develop prognostic and etiologic models for the patients that are most likely to respond to acupuncture. If a clinically important benefit for acupuncture is found, a broader application of this technique would be justified. However, if the results are negative, then the addition of acupuncture to EPT should be generally curtailed.

ELIGIBILITY:
INCLUSION CRITERIA

* X-ray proven osteoarthritis of the knee - Kellgren level 2 or greater
* More than 3 months of moderate knee pain
* Previous trial of NSAIDs or acetaminophen
* Physician referral for at least 6 physical therapy treatments
* Capacity to understand the requirements of the study and complete questionnaires

  * Average knee pain with movement, 4 or above, during the last week

EXCLUSION CRITERIA

* Average hip, back, ankle pain is greater than average knee pain (scale 1-10)
* Back, hip or ankle pain substantially interferes with patient knee assessment
* History of gout

  * Acupuncture in the last year
  * Moderate or greater hip or ankle pain greater than 3 daily
  * Local corticosteroid injection into the effected knee within the past 4 weeks
  * Hyaluronidase within the past 6 months
  * Bleeding disorder or current use of Coumadin or Heparin
  * Cardiac or pulmonary disease limiting exercise tolerance enough to limit the standard exercise physical therapy
  * History of alcohol or drug abuse within the past 6 months
  * Unable to complete a six minute walk test

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2002-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John T. Farrar, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Penn Therapy and Fitness, Philadelphia, Pennsylvania
  - Veterans Administration Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital Sports Medicine/Rehabilitation Center, Philadelphia, Pennsylvania